CLINICAL TRIAL: NCT01682135
Title: Phase I Study of Ramucirumab in Patients With Advanced Solid Tumors
Brief Title: A Study in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14139; I4T-CR-JVBU (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Results first posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-07

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ramucirumab (Experimental): Ramucirumab administered intravenously (IV) at escalating doses (6 milligrams per kilogram [mg/kg] up to 10 mg/kg) every 2-3 weeks for 6 weeks (1 Cycle). Treatment may continue until discontinuation criterion is met.
  Interventions: Biological: Ramucirumab

INTERVENTIONS:
Biological: Ramucirumab — Administered IV.
  Other Names: IMC-1121B; LY3009806

SUMMARY:
This trial is testing ramucirumab (LY3009806) administered to Chinese participants with advanced solid tumors that are resistant to standard therapy or for whom no standard therapy is available. The purpose of this study is to evaluate how safe ramucirumab is and whether it causes any side effects. The study will also measure how much ramucirumab gets into the blood stream and how long it takes the body to get rid of it.

ELIGIBILITY:
Inclusion Criteria:

* Chinese participants with histopathologically or cytologically diagnosed advanced solid tumor
* Did not respond to standard therapy or no standard therapy is available
* Measurable or nonmeasurable disease according to the Response Evaluation Criteria In Solid Tumors (RECIST)
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1 at study entry
* Able to provide written informed consent
* A life expectancy of >3 months
* Adequate hematologic function, as defined by: Absolute neutrophil count (ANC) ≥1500 per cubic millimeter (mm^3); hemoglobin concentration ≥9 grams per deciliter (g/dL); and platelet count ≥100,000/mm^3
* Adequate hepatic function, as defined by: Total bilirubin level ≤1.5 x the upper limit of normal (ULN) (in participants with known Gilbert Syndrome, a total bilirubin ≤ 3.0 x ULN with direct bilirubin ≤ 1.5 x ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x ULN (or ≤5 x ULN if the participant has liver metastases
* Adequate renal function, as defined by: Serum creatinine level ≤1.5 x ULN; or calculated serum creatinine clearance (Cockcroft-Gault) ≥50 milliliters per minute (mL/min)
* Urinary protein is 0 or 1+ on dipstick but no edema nor serum albumin < lower level of normal
* Adequate coagulation function, as defined by: International normalized ratio (INR) ≤1.5, or prothrombin time (PT) ≤1.5 x ULN and activated partial thromboplastin time (aPTT) ≤1.5 x ULN (unless receiving anticoagulation therapy)
* Agrees to use adequate contraception during the study period and for 12 weeks after the last dose of study treatment

Exclusion Criteria:

* Had chemotherapy or therapeutic radiotherapy within 14 days (6 weeks for nitrosoureas or mitomycin C) before entering the study or the participant has ongoing side effects (≥ Grade 2) due to previously administered agents
* Has obvious evidence of intratumor cavitation
* Has undergone major surgery within 28 days before study entry or has had a central venous access device inserted within 7 days before study entry
* Has a history of gastrointestinal perforation, postoperative bleeding complications, or wound complications from a surgical procedure
* Has elective or planned surgery to be conducted during the trial
* Has documented and/or symptomatic brain or leptomeningeal metastases
* Has uncontrolled ongoing illness, for example: thrombotic or hemorrhagic disorders; hemoptysis; ongoing infection requiring systemic antibiotic treatment; congestive heart failure, angina pectoris, angioplasty, stenting, or myocardial infarction within 6 months; stroke, transient ischemic attack (TIA), or other grade 3-4 arterial thromboembolic event occurring within 6 months; uncontrolled hypertension (≥150/≥90 millimeters of mercury [mmHg]); cardiac arrhythmia that requires treatment or asymptomatic sustained ventricular tachycardia; peripheral neuropathy ≥Grade 2; human immunodeficiency virus (HIV) or active, uncontrolled hepatitis, liver cirrhosis at a level of Child-Pugh Class B (or worse), liver cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. (Clinically meaningful ascites is defined as ascites resulting from cirrhosis and requiring ongoing treatment with diuretics and/or paracentesis)
* Has a serious or nonhealing wound, ulcer, or bone fracture within 28 days before study entry
* Has experienced any Grade 3 or 4 gastrointestinal bleeding within 3 months before study entry
* Has a history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess <6 months before randomization, or the participant has a history of poorly controlled or recurrent inflammatory bowel disease (including Crohn's disease or ulcerative colitis)
* Has participated in a clinical study of a non-approved experimental agent or procedure within 4 weeks prior to study entry for small molecules, or 8 weeks before study entry for non-approved monoclonal antibodies
* Has a known allergy to ramucirumab or its excipients, a monoclonal antibody (MAb), or any other therapeutic protein, such as fresh frozen plasma, human serum albumin (HSA), cytokines, or interleukins. If there is suspicion that the participant may have an allergy, the participant should be excluded
* Is pregnant (confirmed by urine or serum pregnancy test) or lactating
* Has known alcohol or drug dependency
* Is receiving chronic therapy with nonsteroidal anti-inflammatory agents (NSAIDs)
* Is not considered to be suitable for this study, in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai, China

REFERENCES:
- [Derived] Cao J, Ji D, Chen Z, Shen W, Wang J, Li B, Chi H, Long A, Gao L, Li J. Phase I Dose-Escalation Study of Ramucirumab in Chinese Patients with Advanced Solid Tumors. Oncologist. 2017 Jun;22(6):638-e56. doi: 10.1634/theoncologist.2017-0137. Epub 2017 May 2. PMID 28465370

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant study completion is defined as a participant either completing all 6 cycles of study drug or discontinuing study drug due to dose-limiting toxicities (DLT), then completing all required End-of-Therapy and End-of-Study assessments.
Groups:
- Cohort 1 - 6 mg/kg/2w Ramucirumab: 6 milligram per kilogram (mg/kg) ramucirumab administered intravenously (IV) every 2 weeks (w) for 6 weeks (one cycle). When a pre-defined percentage of participants completed Cycle 1 without experiencing a DLT, dose escalation was initiated with the start of Cohort 2. After Cycle 1 treatment, participants who had an objective response or stable disease were permitted to receive ramucirumab at the same dose and schedule until disease progression or unacceptable toxicity occurred, or another withdrawal criterion was met.
- Cohort 2 - 10 mg/kg/3w Ramucirumab: 10 mg/kg ramucirumab administered IV every 3 weeks for 6 weeks (one cycle). When a pre-defined percentage of participants completed Cycle 1 without experiencing a DLT, dose escalation was initiated with the start of Cohort 3. After Cycle 1 treatment, participants who had an objective response or stable disease were permitted to receive ramucirumab at the same dose and schedule until disease progression or unacceptable toxicity occurred, or another withdrawal criterion was met.
- Cohort 3 - 8 mg/kg/2w Ramucirumab: 8 mg/kg ramucirumab administered IV every 2 weeks for 6 weeks (one cycle). After Cycle 1 treatment, participants who had an objective response or stable disease were permitted to receive ramucirumab at the same dose and schedule until disease progression or unacceptable toxicity occurred, or another withdrawal criterion was met.
Period: Overall Study
Arm/Group | Cohort 1 - 6 mg/kg/2w Ramucirumab | Cohort 2 - 10 mg/kg/3w Ramucirumab | Cohort 3 - 8 mg/kg/2w Ramucirumab
Started | 6 | 10 | 12
Received at Least 1 Dose of Study Drug | 6 | 10 | 12
Completed | 6 | 10 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Cohort 1 - 6 mg/kg/2w Ramucirumab: 6 mg/kg ramucirumab administered IV every 2 weeks for 6 weeks (one cycle) followed by dose escalation to Cohort 2. When a pre-defined percentage of participants completed Cycle 1 without experiencing a DLT, dose escalation was initiated with the start of Cohort 2.
- Cohort 2 - 10 mg/kg/3w Ramucirumab: 10 mg/kg ramucirumab administered IV every 3 weeks for 6 weeks (one cycle) followed by dose escalation to Cohort 3. When a pre-defined percentage of participants completed Cycle 1 without experiencing a DLT, dose escalation was initiated with the start of Cohort 3.
- Cohort 3 - 8 mg/kg/2w Ramucirumab: 8 mg/kg ramucirumab administered IV every 2 weeks for 6 weeks (one cycle).
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - 6 mg/kg/2w Ramucirumab | Cohort 2 - 10 mg/kg/3w Ramucirumab | Cohort 3 - 8 mg/kg/2w Ramucirumab | Total
Number analyzed (Participants) | 6 | 10 | 12 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.20 (9.060) | 52.92 (9.509) | 58.18 (9.444) | 54.80 (9.536)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7 | 14
  Male | 2 | 7 | 5 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 10 | 12 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  China | 6 | 10 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Drug-Related Adverse Events (AEs) or Any Serious Adverse Events (SAEs)
Description: A summary of AEs and SAEs considered by the investigator to be drug-related is located in the Reported Adverse Events module. An AE is summarized if the onset date is on or after the first dose of study drug and within 30 days after the last dose, or it occurred before the first dose of study drug and worsened while on the therapy.
Time Frame: Baseline through Study Completion (Up to 12 Weeks)
Population: All enrolled participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Groups:
- Cohort 1: 6 mg/kg/2w Ramucirumab: 6 mg/kg ramucirumab administered intravenously (IV) every 2 weeks (w) for 6 weeks (one cycle). When a pre-defined percentage of participants completed Cycle 1 without experiencing a DLT, dose escalation was initiated with the start of Cohort 2.
- Cohort 2: 10 mg/kg/3w Ramucirumab: 10 mg/kg ramucirumab administered IV every 3 weeks for 6 weeks (one cycle). When a pre-defined percentage of participants completed Cycle 1 without experiencing a DLT, dose escalation was initiated with the start of Cohort 3.
- Cohort 3: 8 mg/kg/2w Ramucirumab: 8 mg/kg ramucirumab administered IV every 2 weeks for 6 weeks (one cycle).
Arm/Group | Cohort 1: 6 mg/kg/2w Ramucirumab | Cohort 2: 10 mg/kg/3w Ramucirumab | Cohort 3: 8 mg/kg/2w Ramucirumab
Number analyzed (Participants) | 6 | 10 | 12
Participants
  Drug-Related Adverse Event | 4 | 8 | 10
  Serious Adverse Event | 0 | 1 | 0

2. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of Ramucirumab
Time Frame: Cycle 1 & 2: Predose, End of Infusion, 0.5 hour (h) ,1h, 2h, 4h, 8h, 24h, 48h,72h or 96h, 168h, 264h, and 336h Postdose (and 504h Postdose Cohort 2 only)
Population: All enrolled participants who received at least one dose of study drug and had evaluable Cmax pharmacokinetics (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (µg/mL)
Groups:
- Cohort 1: 6 mg/kg/2w Ramucirumab: 6 mg/kg ramucirumab administered IV every 2 weeks for 6 weeks (one cycle). When a pre-defined percentage of participants completed Cycle 1 without experiencing a DLT, dose escalation was initiated with the start of Cohort 2.
Arm/Group | Cohort 1: 6 mg/kg/2w Ramucirumab | Cohort 2: 10 mg/kg/3w Ramucirumab | Cohort 3: 8 mg/kg/2w Ramucirumab
Number analyzed (Participants) | 6 | 9 | 12
microgram/milliliter (µg/mL)
  Cycle 1 (n = 6, 9, 12) | 155 (13) | 186 (22) | 190 (39)
  Cycle 2 (n = 1, 6, 8) | NA (NA) — Geometric Mean and %CV not calculated for 1 participant. Individual Value = 155 µg/mL. | 219 (22) | 239 (19)

3. Primary Outcome: Pharmacokinetics: Minimum Concentration (Cmin) of Ramucirumab
Time Frame: Cycle 2-5: Predose
Population: All enrolled participants who received at least one dose of study drug and had evaluable Cmin PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Cohort 1: 6 mg/kg/2w Ramucirumab | Cohort 2: 10 mg/kg/3w Ramucirumab | Cohort 3: 8 mg/kg/2w Ramucirumab
Number analyzed (Participants) | 5 | 8 | 10
µg/mL
  Cycle 2 (n = 5, 8, 10) | 36.9 (35) | 29.5 (90) | 59.7 (26)
  Cycle 3 (n = 1, 2, 5) | NA (NA) — Geometric Mean and %CV not calculated for 1 participant. Individual Value = 37.1 µg/mL. | NA (NA) — Geometric Mean and %CV not calculated for 2 participants. Individual Values = 41.2 and 50.2 µg/mL. | 68.7 (28)
  Cycle 4 (n = 1, 2, 4) | NA (NA) — Geometric Mean and %CV not calculated for 1 participant. Individual Value = 51.9 µg/mL. | NA (NA) — Geometric Mean and %CV not calculated for 2 participants. Individual Values = 56.0 and 84.1 µg/mL. | 79.6 (26)
  Cycle 5 (n = 0, 3, 4) | NA (NA) — Geometric Mean and %CV not calculated for 0 participants; no data. | 56.5 (17) | 92.5 (19)

4. Primary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve (AUC) of Ramucirumab
Description: Cycle 1 analysis performed: Area Under the Concentration-Time Curve Zero to Infinity (AUC[0-∞]); Cycle 2 analysis performed: Area Under the Concentration-Time Curve Over the Dosing Interval at Steady State (AUC[τ,ss])
Time Frame: as for outcome 2
Population: All enrolled participants who received at least one dose of study drug and had evaluable AUC(0-∞) for Cycle 1 and AUC(τ,ss) for Cycle 2 PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*day/milliliter (µg*day/mL)
Arm/Group | Cohort 1: 6 mg/kg/2w Ramucirumab | Cohort 2: 10 mg/kg/3w Ramucirumab | Cohort 3: 8 mg/kg/2w Ramucirumab
Number analyzed (Participants) | 5 | 7 | 7
Microgram*day/milliliter (µg*day/mL)
  Cycle 1 AUC(0-∞) (n = 5, 7, 7) | 870 (14) | 1430 (31) | 1350 (9)
  Cycle 2 AUC(τ,ss) (n = 1, 6, 8) | NA (NA) — Geometric Mean and %CV not calculated for 1 participant. Mean Value = 892 µg*day/mL). | 1630 (32) | 1540 (16)

5. Secondary Outcome: Duration of Response
Description: Participants achieved an objective response if they had a best overall response of complete response (CR) or partial response (PR). According to RECIST v1.1, CR was the disappearance of all non-nodal target lesions, with the short axes of any target lymph node reduced to <10 mm, the disappearance of all nontarget lesions, and the normalization of tumor marker levels (if tumor markers were initially above the upper limit of normal); PR was defined as at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph node), taking as reference the baseline sum diameter. For each participant who is not known to have died or to have had objective progression of disease as of the data-inclusion cut-off date for a particular analysis, duration of tumor response was to be censored at the date of the participant's last objective tumor assessment prior to that cut-off date.
Time Frame: Time Between Meeting Response Criteria and Progressive Disease or Death Due to Any Cause (Up to 10 Weeks)
Population: All enrolled participants who received at least one dose of study drug. There were no participants censored due to no CR or PR responses.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: 6 mg/kg/2w Ramucirumab | Cohort 2: 10 mg/kg/3w Ramucirumab | Cohort 3: 8 mg/kg/2w Ramucirumab
Number analyzed (Participants) | 6 | 10 | 12
Months | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

6. Secondary Outcome: Duration of Stable Disease (SD)
Description: Duration of SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum of diameters while on study. SD is measured at the start of the study drug until progressive disease or death due to any cause, whichever is first. Censoring occurred if a participant did not have a complete baseline disease assessment, initiated on another anti-cancer therapy (censored at the date of the last complete objective progression-free disease assessment before initiation of the new therapy), was not known to have died or had objective progression as of the data inclusion cutoff date for analysis.
Time Frame: Baseline to Progressive Disease or Death Due to Any Cause (Up to 10 Weeks)
Population: All enrolled participants who received at least one dose of study drug and had evaluable SD data. Participants censored for Cohort 1, 2, and 3: 3, 2, and 1, respectively.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: 6 mg/kg/2w Ramucirumab | Cohort 2: 10 mg/kg/3w Ramucirumab | Cohort 3: 8 mg/kg/2w Ramucirumab
Number analyzed (Participants) | 3 | 7 | 8
Months | NA [NA to NA] — The number of values in this cohort was too small to calculate due to censoring. | 5.68 [2.79 to 12.22] | 5.29 [2.92 to 6.87]

7. Secondary Outcome: Time to Disease Progression
Description: Time to progressive disease was measured from the start of study drug until progressive disease. Censoring occurred if a participant did not have a complete baseline disease assessment, initiated on another anti-cancer therapy (censored at the date of the last complete objective progression-free disease assessment before initiation of the new therapy), was not known to have died or had objective progression as of the data inclusion cutoff date for analysis.
Time Frame: Baseline to Progressive Disease (Up to 10 Weeks)
Population: All enrolled participants who received at least one dose of study drug. Censoring for Cohort 1, 2 and 3: 3, 2 and 2, respectively.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Cohort 3: 8 mg/kg/2w Ramucirumab: 8mg/kg ramucirumab administered IV every 2 weeks for 6 weeks (one cycle).
Arm/Group | Cohort 1: 6 mg/kg/2w Ramucirumab | Cohort 2: 10 mg/kg/3w Ramucirumab | Cohort 3: 8 mg/kg/2w Ramucirumab
Number analyzed (Participants) | 6 | 10 | 12
Months | 1.41 [1.35 to NA] — The number of values in this cohort was too small to calculate due to censoring. | 3.38 [1.28 to 8.21] | 3.94 [1.22 to 5.55]

8. Secondary Outcome: Number of Participants With Anti-Ramucirumab Antibodies
Description: A sample will be considered positive for circulating anti-ramucirumab antibodies if it exhibits a post-baseline antibody level that exceeds the upper 95% confidence interval of the mean determined from the normal anti-ramucirumab level seen in healthy untreated individuals. A participant will be considered to have an anti-ramucirumab response if there are 2 consecutive positive samples or if the final sample tested is positive.
Time Frame: Cycle 1: Pre-infusion, Cycle 2: Pre-infusion, Cycle 3: Pre-infusion
Population: All enrolled participants who received at least one dose of study drug and had evaluable immunogenicity data.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: 6 mg/kg/2w Ramucirumab | Cohort 2: 10 mg/kg/3w Ramucirumab | Cohort 3: 8 mg/kg/2w Ramucirumab
Number analyzed (Participants) | 6 | 10 | 12
Participants | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Best Objective Response (BOR)
Description: Participants achieved disease control if they had a BOR of CR, PR or SD. Progressive Disease (PD) and those participants which were Not Evaluable (NE) were also reported. According to RECIST v1.1, CR was the disappearance of all non-nodal target lesions, with the short axes of any target lymph node reduced to <10 mm, the disappearance of all nontarget lesions, and the normalization of tumor marker levels (if tumor markers were initially above the upper limit of normal); PR was defined as at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph node), taking as reference the baseline sum diameter. SD was neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD, taking as reference the smallest sum diameter since treatment started.
Time Frame: Baseline to Progressive Disease or Participant Stopped Study (Up to 10 Weeks)
Population: All enrolled participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: 6 mg/kg/2w Ramucirumab | Cohort 2: 10 mg/kg/3w Ramucirumab | Cohort 3: 8 mg/kg/2w Ramucirumab
Number analyzed (Participants) | 6 | 10 | 12
Participants
  Complete Response (CR) | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 0
  Stable Disease (SD) | 3 | 7 | 8
  Progressive Disease (PD) | 3 | 3 | 3
  Not Evaluable (NE) | 0 | 0 | 1

ADVERSE EVENTS:
Groups:
- Cohort 1 - 6mg/kg/2w Ramucirumab: 6mg/kg ramucirumab administered IV every 2 weeks for 6 weeks (one cycle). When a pre-defined percentage of participants completed Cycle 1 without experiencing a DLT, dose escalation was initiated with the start of Cohort 2.
- Cohort 2 - 10mg/kg/3w Ramucirumab: 10mg/kg ramucirumab administered IV every 3 weeks for 6 weeks (one cycle). When a pre-defined percentage of participants completed Cycle 1 without experiencing a DLT, dose escalation was initiated with the start of Cohort 3.
- Cohort 3 - 8mg/kg/2w Ramucirumab: 8mg/kg ramucirumab administered IV every 2 weeks for 6 weeks (one cycle).
Arm/Group | Cohort 1 - 6mg/kg/2w Ramucirumab | Cohort 2 - 10mg/kg/3w Ramucirumab | Cohort 3 - 8mg/kg/2w Ramucirumab
Serious Adverse Events (participants affected / at risk) | 1/6 | 2/10 | 1/12
Other Adverse Events (participants affected / at risk) | 6/6 | 10/10 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 6mg/kg/2w Ramucirumab (N=6) | Cohort 2 - 10mg/kg/3w Ramucirumab (N=10) | Cohort 3 - 8mg/kg/2w Ramucirumab (N=12)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort 1 - 6mg/kg/2w Ramucirumab (N=6) | Cohort 2 - 10mg/kg/3w Ramucirumab (N=10) | Cohort 3 - 8mg/kg/2w Ramucirumab (N=12)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 1 (2) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 3 (27) | 4 (10)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (4) | 1 (1) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 3 (8)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (3)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 4 (9) | 2 (3)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 2 (2) | 1 (1) | 2 (2)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 6 (8) | 8 (11) | 5 (5)
Influenza like illness (General disorders) | 0 (0) | 2 (2) | 3 (4)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 4 (5)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 2 (2)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0/4 (0) | 1/3 (1) | 0/7 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 5 (9) | 5 (11)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 5 (8) | 7 (13)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram st segment abnormal (Investigations) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram t wave abnormal (Investigations) | 0 (0) | 3 (5) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Glucose urine present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 4 (8) | 1 (1)
Platelet count decreased (Investigations) | 1 (2) | 4 (4) | 1 (2)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 2 (2) | 3 (4)
White blood cell count decreased (Investigations) | 2 (3) | 3 (7) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 3 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2) | 3 (3) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 3 (5) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 3 (4)
Headache (Nervous system disorders) | 1 (2) | 2 (3) | 4 (7)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 3 (8) | 3 (5) | 6 (8)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0/4 (0) | 1/3 (2) | 0/7 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (6) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 3 (8) | 7 (29) | 5 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days